CLINICAL TRIAL: NCT02768038
Title: The Role of Intestinal Microbiome ih the Pathogenesis and Course of Chronic Inflammatory Bowel Diseases
Brief Title: Intestinal Microbiome and Chronic Inflammatory Bowel Disease
Status: Withdrawn | Type: Observational
Why Stopped: The researcher (Ph student) interrupted the dissertation project
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TurkuUH2
Record Dates: First submitted 2015-12-16; First posted 2016-05-11 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Colitis
MeSH Terms: conditions — Colitis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood and stool specimens. Biopsy specimens from large intestine ja ileum.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational — Blood, stool ja biopsy specimens

SUMMARY:
The aim is to examine the role of intestinal microbiota in the pathogenesis of chronic inflammatory bowel diseases (IBD)

DETAILED DESCRIPTION:
IBD patients to whom colonoscopy is performed will be recruited. Mucosal specimens from large intestine and terminal ileum will be collected as well as stool specimens. The microbiota will be analyzed at the microbiology laboratory and the results will be correlated with endoscopical, laboratory and histopathological findings.

ELIGIBILITY:
Inclusion Criteria:

* IBD

Exclusion Criteria:

* patient refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBD living at the Turku University Hospital area
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of microbiome in chronic inflammatory bowel disease | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Markku Voutilainen, Prof., Principal Investigator — Head, Department of Gastroenterology
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No